CLINICAL TRIAL: NCT04168255
Title: Perfluorocarbone Liquids for Tamponading Lower Retinal Breaks to Achieve Retinal Reattachment in Eyes of Retinal Detachment With Proliferative Vitreoretinopathy
Brief Title: Double Retinal Tamponade for Retinal Detachment With PVR and Inferior Breaks.
Acronym: IRB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Shaaban Elwan, Assistant professor of ophthalmology, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Minia University,IRB
Record Dates: First submitted 2019-11-16; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Intervention Model Description: Retinal detachment with proliferative vitreoretinopathy and inferior breaks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Retinal detachment (Other): Retinal detachment with proliferative vitreoretinopathy and inferior breaks
  Interventions: Procedure: Double tamponade

INTERVENTIONS:
Procedure: Double tamponade — Double tamponade procedure in retinal detachment with PVR and inferior breaks

SUMMARY:
Purpose To evaluate the efficacy of perfluorocarbone liquids (PFCLs) for tamponading lower retinal breaks to achieve retinal reattachment in eyes of retinal detachment with proliferative vitreoretinopathy (PVR) and inferior breaks.

Patients and methods The study was prospective non comparative interventional study. It included thirty eyes of 30 patients suffering from retinal detachment with proliferative vitreoretinopathy and inferior breaks attending the ophthalmology department at Minia University Hospital. The mean age was 50.2± 10.63 years, 18 females and 12 males. Double retinal tamponade procedure were done and the patients were followed for one year. The primary outcome was to achieve successful retinal reattachment and the secondary outcome is to achieve improvement in the postoperative visual acuity.

DETAILED DESCRIPTION:
Patients and methods The study includes thirty eyes of 30 patients with dense cataract, retinal detachment (RD) and proliferative vitreoretinopathy (PVR) and inferior breaks (18 females and 12 males) in the period from October, 2017 to August, 2019 at ophthalmology department, Minia University Hospital. Approval of the study was provided by Faculty of Medicine, Research Ethics Committee and it was in agreement with the tents of Declaration of Helsinki and all patients were singed a consent explaining the risk and benefits of their operation. All of the patients was followed for 12 months.

Preoperative examinations History taking included age, sex, laterality and systemic diseases and medications. Ophthalmological examinations including visual acuity assessment, IOP measurement, anterior segment slit lamp examinations, Dilated fundus examinations using indirect ophthalmoscope as well as with the auxiliary lenses and slit lamp aid, retinal chart drawing, biometry and ultrasonography if needed.

Surgical technique All of cases were done under peribulbar anesthesia. First, phacoemulsification was performed through clear corneal temporal incision with implantation of hydrophobic acrylic IOL in the capsular bag and closure of wound by a 10/0 nylon suture. This was followed by 23-G pars plana vitrectomy. Core vitrectomy was done and triamcinolone acetonide was injected to ensure complete posterior vitreous detachment. All epiretinal membranes were removed helped by the use of membrane blue (trypan blue 0.15%, DORC International). Then, perfluorocarbone liquid (PFCL) was injected to flatten the posterior retina and base vitrectomy was performed helped by scleral depression. More PFCL was injected to drain subretinal fluid through the original retinal breaks. All retinal breaks were surrounded by 3-4 rows of diode endolaser photocoagulation. Then, fluid air exchange was performed to aspirate PFCL leaving a part of it enough to tamponade the lower retinal breaks and 12% C3F8 (perfluoropropane) was injected into the eye. After 2 weeks, the remaining PFCL was aspirated and replaced with 12% C3F8.

Post-operative management All patients were given topical prednisolone 1% (Optipred, Jamjoom pharma Co.) eye drops (QID) and tapered through 4-6 weeks, cyclopentolate 0.5 % eye drops (TID), moxifloxacin 0.3 mg (Vigamox, Alcon Co.) eye drops QID for 1 week and Maxitrol ointment (Neomycin sulphate 3.5 mg, Polymyxin B sulphate 10000 IU and dexamethasone 0.1%, Alcon Co) at night for 4 weeks. Follow up visits were advised next postoperative day, one week, , one month, and then each three months for 1 year.

All patients underwent full ophthalmologic examination including BCDVA, IOP, anterior segment slit lamp examination, and dilated fundus examination. Baseline results and that of 1, 3 6, 9 months, and 1year were included in the statistical analysis. This study primary outcome is to achieve successful retinal reattachment and the secondary outcome is to achieve improvement in the visual acuity (BCDVA, log MAR). Successful surgery was considered when retinal reattachment was achieved, improvement in the visual acuity without serious complications such as suprachoroidal hemorrhage, retinal detachment or endophthalmitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients had retinal detachment with mild to moderate PVR and inferior retinal breaks fit for the operation and patients that completed all the required follow up visits.

Exclusion Criteria:

* Rhegmatogenous retinal detachment without inferior breaks, other causes of retinal detachment; (tractional or exudative), cases of severe PVR and closed funnel, retinal vascular disorders, maculopathies, uveitis, glaucoma, corneal opacities and previous retinal re-attachment surgery.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
retinal reattachment | one year
  to achieve successful retinal reattachment

SECONDARY OUTCOMES:
visual acuity | 1 year
  is to achieve improvement in the visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Shaaban A Elwan, MD, Principal Investigator — Minia University
Locations (1):
- Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
methdology
Supporting Information: CSR
Time Frame: soon and for 2 years
Access Criteria: Methdology

REFERENCES:
- [Background] Yu Q, Liu K, Su L, Xia X, Xu X. Perfluorocarbon liquid: its application in vitreoretinal surgery and related ocular inflammation. Biomed Res Int. 2014;2014:250323. doi: 10.1155/2014/250323. Epub 2014 Mar 30. PMID 24800216
- [Derived] Farouk Abdelkader M, Abd-Elhamid Mehany Elwan S, Shawkat Abdelhalim A. Double Retinal Tamponade for Treatment of Rhegmatogenous Retinal Detachment with Proliferative Vitreoretinopathy and Inferior Breaks. J Ophthalmol. 2020 Oct 7;2020:6938627. doi: 10.1155/2020/6938627. eCollection 2020. PMID 33083050